CLINICAL TRIAL: NCT01420614
Title: RadIal Versus Femoral Randomized InvEstigation in ST Elevation Acute Coronary Syndrome
Brief Title: RadIal Versus Femoral InvEstigation in ST Elevation Acute Coronary Syndrome
Acronym: RIFLE-STEACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Policlinico Casilino ASL RMB (Other)
Responsible Party: Principal Investigator, Enrico Romagnoli, MD, PhD, Policlinico Casilino ASL RMB
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PC-03ER
Record Dates: First submitted 2011-08-15; First posted 2011-08-19 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome; ST Elevation Acute Myocardial Infarction
Keywords: radial access; primary angioplasty; trial; randomization; outcome
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radial (Experimental): group of patients undergoing primary angioplasty by transradial approach
  Interventions: Procedure: Radial approach
- Femoral (Active Comparator): group of patients undergoing primary angioplasty by transfemoral approach
  Interventions: Procedure: Femoral approach

INTERVENTIONS:
Procedure: Femoral approach — diagnostic and interventional procedures by femoral artery access
  Other Names: transfemoral
  Arms: Femoral
Procedure: Radial approach — diagnostic and interventional procedures by radial artery access
  Other Names: transradial
  Arms: Radial

SUMMARY:
Prospective, randomized, multi-center trial comparing the safety and efficacy in the prevention of net adverse clinical outcomes (NACE) of transfemoral vs. transradial approach for the treatment of patients with ST-elevation acute coronary syndrome (STEACS) undergoing primary angioplasty

DETAILED DESCRIPTION:
Prospective, randomized, double arm study. The study population will include all consecutive patients presenting with a ST-elevation Acute Coronary Syndrome and candidates for primary percutaneous coronary intervention, who agree and provide written informed consent for the study.

Before arterial stick for percutaneous access, patients will be randomized according to sealed numbered envelopes. Subsequently, arterial access will be obtained and the diagnostic/interventional procedure will be performed according to routine clinical practice, leaving ancillary medications, choice of devices and means of hemostasis at the physician's discretion.

In the randomization process all participating centers will be equally stratified to avoid statistical unbalance.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is >18 years old with recent acute ST-elevation acute coronary syndrome (STEACS) requiring emergent coronary angiography.
2. Patient has no contraindication to percutaneous arterial access by both and transfemoral route.
3. Subject has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee of the respective clinical site.
4. Patient and the treating physician agree that the subject will comply with all follow-up evaluations.

Exclusion Criteria:

1. Subject's age is <18 years and he has no acute ST-elevation myocardial infarction (ST elevation of a least 0.1 mV in ≥2 extremity leads or at least 0.2 mV in ≥2 precordial leads).
2. Subject has had a recent stroke or TIA (<4 weeks), irrespective of age.
3. Patient has an international normalized ratio (INR) > 2.0, or other severe bleeding diathesis
4. The patient is pregnant or breastfeeding.
5. Known allergies to: aspirin, clopidogrel and ticlopidine, heparin, IIb/IIIa inhibitors, stainless steel, or contrast agent (which cannot be adequately premedicated).

7.Subject is currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints.

8.Prior participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1001 (Actual)
Dates: Start 2009-01; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Net Adverse Clinical Event | 30-day
  Cumulative of cardiac death, myocardial infarction, target lesion revascularization, stroke and bleeding

SECONDARY OUTCOMES:
Net Adverse Clinical Event | 1-year
  Cumulative of cardiac death, myocardial infarction, target lesion revascularization, stroke and bleeding
Individual components of NACE | 30-day
  Cardiac death, Myocardial infarction, Target Lesion revascularization, Stroke, Major Bleeding
Individual components of NACE | 1-year
  Cardiac death, Myocardial infarction, Target Lesion revascularization, Stroke, Major Bleeding
Total procedural and fluoroscopy times for the index procedure | 1 day
  Comparison of procedural and fluoroscopy times between the two study groups
Hospital stay | 30-day
  Days of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Lioy, MD, Principal Investigator — Policlinico Casilino
Locations (4):
- Italy (4):
  - Università di Modena e Reggio Emilia, Modena, Modena
  - Ospedale Sandro Pertini, Rome, Rome
  - Policlinico Casilino, Rome, Rome
  - University of Turin, San Giovanni Battista Hospital, Turin, Turin

REFERENCES:
- [Derived] Romagnoli E, Biondi-Zoccai G, Sciahbasi A, Politi L, Rigattieri S, Pendenza G, Summaria F, Patrizi R, Borghi A, Di Russo C, Moretti C, Agostoni P, Loschiavo P, Lioy E, Sheiban I, Sangiorgi G. Radial versus femoral randomized investigation in ST-segment elevation acute coronary syndrome: the RIFLE-STEACS (Radial Versus Femoral Randomized Investigation in ST-Elevation Acute Coronary Syndrome) study. J Am Coll Cardiol. 2012 Dec 18;60(24):2481-9. doi: 10.1016/j.jacc.2012.06.017. Epub 2012 Aug 1. PMID 22858390